CLINICAL TRIAL: NCT03059940
Title: Optimizing Effectiveness of Smoking Cessation Intervention During Low Dose CT Screening for Lung Cancer
Brief Title: Smoking Cessation Intervention During Low Dose CT (LDCT) Screening for Lung Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0626; R01-CA 2027078-01 (Other Grant/Funding Number: NCI); NCI-2018-01219 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Low Dose computed tomography; LDCT; Quitline; Questionnaires; Surveys; Counseling; Smoking cessation drugs; Anti-Smoking Drug; Nicotine replacement therapy; NRT; Nicotine Patch
MeSH Terms: conditions — Smoking Cessation | interventions — Surveys and Questionnaires; Videotape Recording; Tobacco Use Cessation Devices; thiamine triphosphorate; Carbon Monoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Quitline (QL) Group (Experimental): Questionnaires completed at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan. CO level measured at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan.
  Participants have a CT scan of chest to look for signs of lung cancer. Participants watch a short video about lung cancer, CT scans, and smoking cessation. Brief cessation counseling given by LDCT provider. Participants given shared decision making and discussion about screening with the LDCT provider.
  Participants referred to the Quitline for counseling and NRT (nicotine patch). Participants have 5 smoking cessation counseling sessions over the next 12 weeks.
  Interventions: Behavioral: Questionnaires; Procedure: Low Dose Computed Tomography Scan; Other: Shared Decision Making + Video; Behavioral: Cessation Counseling; Behavioral: Quitline; Drug: Nicotine Patch; Other: Carbon Monoxide (CO) Level Test
- Quitline-Rx (QL-Rx) Group (Experimental): Questionnaires completed at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan. CO level measured at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan.
  Participants have a CT scan of chest to look for signs of lung cancer. Participants watch a short video about lung cancer, CT scans, and smoking cessation. Brief cessation counseling given by LDCT provider.
  LDCT provider and patient discuss options for pharmacotherapy.
  Participants referred to the Quitline for counseling. Participants have 5 smoking cessation counseling sessions over the next 12 weeks.
  Interventions: Behavioral: Questionnaires; Procedure: Low Dose Computed Tomography Scan; Other: Shared Decision Making + Video; Behavioral: Cessation Counseling; Behavioral: Quitline; Behavioral: Pharmacotherapy Discussion; Drug: Anti-Smoking Drug; Other: Carbon Monoxide (CO) Level Test
- Integrated Care (IC) Group (Experimental): Questionnaires completed at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan. CO level measured at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan.
  Participants have a CT scan of chest to look for signs of lung cancer. Participants watch a short video about lung cancer, CT scans, and smoking cessation. Brief cessation counseling given by LDCT provider.
  Participant referred to Tobacco Treatment Program (TTP). TTP provides 4-8 counseling sessions and pharmacotherapy over a 10-12 week period,
  Interventions: Behavioral: Questionnaires; Procedure: Low Dose Computed Tomography Scan; Other: Shared Decision Making + Video; Behavioral: Cessation Counseling; Behavioral: Pharmacotherapy Discussion; Drug: Anti-Smoking Drug; Behavioral: Tobacco Treatment Program; Other: Carbon Monoxide (CO) Level Test

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires completed at baseline and at 6 weeks, 12 weeks, and 6 months after the CT scan.
  Other Names: Surveys
Procedure: Low Dose Computed Tomography Scan — Participants have a CT scan of chest to look for signs of lung cancer.
  Other Names: LDCT
Other: Shared Decision Making + Video — Participants given shared decision making and discussion about screening with the LDCT provider. Participants watch a short video about lung cancer, CT scans, and smoking cessation.
Behavioral: Cessation Counseling — Brief cessation counseling given by LDCT provider.
Behavioral: Quitline — Participants referred to the Quitline for counseling. Participants have 5 smoking cessation counseling sessions over the next 12 weeks.
  Arms: Quitline (QL) Group; Quitline-Rx (QL-Rx) Group
Behavioral: Pharmacotherapy Discussion — Participant informed of the risk, benefits and relative efficacy of cessation medications and to assess their medication preferences, expectations and medical suitability for either option. At the conclusion of this conversation the patient is provided with an initial supply of the medication jointly decided between provider and patient.
  Arms: Integrated Care (IC) Group; Quitline-Rx (QL-Rx) Group
Drug: Nicotine Patch — Nicotine patch dispensed. Dosing at physician's discretion.
  Arms: Quitline (QL) Group
Drug: Anti-Smoking Drug — Varenicline or Buproprion prescribed by study doctor with directions of when and how much of anti-smoking drug that should be taken each time.
  Arms: Integrated Care (IC) Group; Quitline-Rx (QL-Rx) Group
Behavioral: Tobacco Treatment Program — Participant referred to Tobacco Treatment Program (TTP). TTP provides 4-8 counseling sessions and pharmacotherapy over a 10-12 week period,
  Other Names: TTP
  Arms: Integrated Care (IC) Group
Other: Carbon Monoxide (CO) Level Test — Participant asked to blow air through a CO-measuring device.
  Other Names: CO

SUMMARY:
The goal of this clinical research study is to offer lung cancer screenings to smokers who want to change their smoking behaviors. All eligible participants will receive smoking cessation counseling and may be offered at least one form of smoking cessation drug. Different forms of counseling (the delivery of counseling and access to counseling) will be compared.

This is an investigational study. Participants on this study will not be prescribed smoking drugs directly by the study staff. However, participants in this study may or may not receive smoking cessation drugs, depending on what the provider thinks is in the participants best interest. All smoking cessation drugs being used are FDA approved and commercially available. It is investigational to compare the different forms of counseling participants receive.

Up to 1260 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will have a CT scan of your chest to look for signs of lung cancer. You will receive the results 0-4 days after the scan. If there are any abnormal areas, you will be referred to your regular doctor for follow-up. No matter what the results are, you will be advised to quit smoking. If you have previously had a low dose CT scan for lung cancer screening in the last 30 days, you may still be eligible to participate in this study. You will be asked to provide documentation of the CT scan results.

You will receive a referral for counseling to help you reduce/quit smoking. You may also discuss medications you can take to reduce smoking.

As part of your counseling treatment, you may be prescribed an FDA-approved and commercially available anti-smoking drug. This may be either nicotine replacement therapy (such as a patch, gum, or lozenge) or an oral drug (such as varenicline or buproprion). The provider will tell you when and how much of your anti-smoking drug you should take each time, based on a discussion between you and your provider. Receiving anti-smoking medication will be done through your counseling treatment and not as part of your participation in this study.

You will have at least 5, but no more than 8, smoking cessation counseling sessions over the next 12 weeks. Each session will last between 30 - 60 minutes, in which you will set a quit date, prepare for your quit date, and discuss coping skills for dealing with smoking "triggers" after your quit date. You will also discuss challenges you may have with quitting.

Study Visits:

You will have 3 additional study visits, at around 6 weeks, 12 weeks, and 6 months after the screening visit, as well as 1 follow-up phone call. At all study visits:

* You will complete questionnaires about several topics, including depression, suicide, and your smoking behavior. These questionnaires should take about 30-45 minutes in total to complete.
* Your CO level will be measured.
* Urine and/or saliva may be collected (at 12 weeks and 6 months only) for a routine test to check your cotinine and nicotine. Cotinine is a chemical released in your body when it breaks down nicotine and will show whether and how much you have recently smoked.

Follow-Up:

About 5 months after you start receiving counseling sessions, you will be called by a member of the study staff and asked about your recent smoking behaviors and habits. This call should last about 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 or older
* Meets guidelines for lung cancer screening, as determined by radiology team
* Reports being a daily or non-daily smoker (any self-reported smoking in the past 30days) and is interested in treatment that might change smoking behavior.
* Able to follow verbal and written instructions in English and complete all aspects ofthe study.
* Provide informed consent and agree to all assessments and study procedures.
* Have an address where he/she can receive mail
* If opting to participate in telemedicine visits, must have a device available to conduct telehealth visits (e.g., smartphone, computer, tablet, etc.).
* Be the only participant in his/her household on active treatment in Protocol 2016-0626at the time.
* Willing and able to undergo low dose CT scan, as determined by radiology team, and has either had a lung cancer screen within 30 days prior to enrollment into this protocol or schedules a LDCT scan for lung cancer screening to occur while taking part in the 2016-0626 protocol.

Exclusion Criteria:

* Current enrollment or plans to enroll in another smoking cessation program in the next6 months.
* Unwilling to refrain from other nicotine substitutes use (i.e., OTC orprescription medication for smoking cessation) or smoking cessation treatments during the course of the the active treatment portion of the study other than what is provided to or recommended for use.
* Current use of certain medications: (1) Smoking cessation meds (last 7 days), that are being used as part of a current attempt to quit smoking i.e., Wellbutrin, Bupropion, Zyban, NRT, Chantix.
* Being pregnant, engaging in breast-feeding, or being of childbearing potential and engaging in sexual activity that could lead to pregnancy and is not protected by a medically acceptable, effective method of birth control while enrolled in the study, as determined by self-report..Medically acceptable contraceptives include: (1) approved hormonal contraceptives (such asbirth control pills, patches, implants or injections), (2) barrier methods (such as a condomor diaphragm) used with a spermicide, or (3) an intrauterine device (IUD).Contraceptive measures sold for emergency use after unprotected sex are not acceptable methodsfor routine use.
* Exclusive use of tobacco products other than cigarettes or little cigars, such as (but not limited to) cigars, chew, snuff, pipe or e-cigs.
* Individuals who are considered clinically unstable and/or unsuitable to participate as determined by the Principal Investigator and/or study physician

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence Rate | 6 months
  Statistical power will focus on primary objective. Primary analyses use intention-to-treat (ITT) principles, with missing observations imputed as smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Robinson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cinciripini PM, Minnix JA, Kypriotakis G, Erasmus J, Beneventi D, Karam-Hage M, Carpenter K, Volk RJ, Carter B, Godoy MCB, Strange C, Shih YT, Cui Y, Green CE, Robinson JD. Smoking Cessation Interventions in the Lung Cancer Screening Setting: A Randomized Clinical Trial. JAMA Intern Med. 2025 Mar 1;185(3):284-291. doi: 10.1001/jamainternmed.2024.7288. PMID 39804633
- See also: MD Anderson Cancer Center — http://www.mdanderson.org